CLINICAL TRIAL: NCT06104033
Title: Practice Change With Drug-coated Balloon in Patients With multiVessel Coronary Artery Disease
Acronym: DCB-MVD
Status: Recruiting | Type: Observational
Sponsor: Bon-Kwon Koo (Other)
Collaborators: Seoul National University Hospital (Other); St Vincent's Hospital (Other); Uijeongbu St. Mary Hospital (Other); Gachon University Gil Medical Center (Other); Gangnam Severance Hospital (Other); Kyunghee University Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Inje University Ilsan Paik Hospital (Other); Daegu Catholic University Medical Center (Other); Sejong General Hospital (Other); Seoul National University Bundang Hospital (Other); Soonchunhyang University Hospital (Other); Yeungnam University Hospital (Other); Wonju Severance Christian Hospital (Other); Ulsan University Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Inje University (Other); Chonnam National University Hospital (Other); Chung-Ang University Gwangmyeong Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Ulsan Medical Center (Other); Hanyang University Seoul Hospital (Other); Jeju National University Hospital (Other); KangWon National University Hospital (Other); Uijeongbu Eulji Medical Center, Eulji University (Unknown); Seoul St. Mary's Hospital (Other); Gyeongsang National University Hospital (Other); Severance Hospital (Other); Chosun University Hospital (Other); Kyungpook National University Hospital (Other); Korea University Anam Hospital (Other); Kyung Hee University Hospital at Gangdong (Other); Ajou University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: 2306-138-1440
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Multi Vessel Coronary Artery Disease
Keywords: Coronary artery disease; Multivessel coronary artery disease; Percutaneous coronary intervention; Drug-coated balloon; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hybrid strategy: The patient undergoes percutaneous coronary intervention with drug-coated balloons and drug-eluting stents or drug-coated balloons only in the coronary artery lesion.
  Interventions: Device: drug-coated balloon; Device: drug-eluting stent
- DES only: The patient undergoes percutaneous coronary intervention with drug-eluting stents only in the coronary artery lesion.
  Interventions: Device: drug-eluting stent

INTERVENTIONS:
Device: drug-coated balloon — For the procedure, the drug-coated balloon (Agent®, Boston Scientific, USA) that can be used for both de-novo coronary lesions and in-stent restenosis lesions is used.
  Groups: Hybrid strategy
Device: drug-eluting stent — When using drug-eluting stents, the latest 2nd generation drug-eluting stent (Synergy®, Boston Scientific, USA) should be used in accordance with the latest guidelines.

SUMMARY:
This study is a prospective, multicenter, open-label, observational study to investigate the impact of using drug-coated balloons (DCBs) in the treatment of coronary artery lesions in patients with multivessel coronary artery disease (MVD), as opposed to the default strategy of using only drug-eluting stents (DES). The investigators aim to assess changes in clinical practice towards a hybrid treatment strategy (DES and DCB) and its effects on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 or older
2. Multivessel coronary artery disease patients requiring coronary intervention

   * Stenosis of 2 or more major coronary arteries or major coronary artery branches (Vessel size ≥2.5mm) with diameter stenosis ≥50% or fractional flow reserve ≤0.80 requiring repeat revascularization
   * Having stenotic lesions requiring revascularization with a vessel size of 2.5mm to 3.0mm
3. Capable of understanding the risks and benefits of participating in the study and providing informed consent

Exclusion Criteria:

1. Incapable of voluntarily providing informed consent
2. Allergy or contraindication to aspirin, P2Y12 inhibitors, or components of drug-eluting stents
3. Cardiogenic shock or cardiac arrest patients
4. Patients with severe left ventricular systolic dysfunction (ejection fraction <30%)
5. Patients for whom coronary artery bypass surgery is prioritized over coronary artery intervention
6. Patients with severe valvular heart disease requiring open heart surgery
7. Pregnant or lactating women

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multivessel coronary artery disease who undergo coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The reclassification rate of the treatment strategy | At the time of procedure
  The reclassification rate according to the change in treatment approach from the default strategy of using only drug-eluting stents (DES-only) to the hybrid strategy of using both drug-coated balloons and drug-eluting stents in the treatment of multivessel coronary artery disease.

SECONDARY OUTCOMES:
Rate of change in treatment pattern from drug-eluting stents to drug-coated balloons in target vessel therapy | At the time of procedure
  Rate of change in treatment pattern from drug-eluting stents to drug-coated balloons in target vessel therapy
Rate of change in treatment pattern from drug-eluting stents to drug-coated balloons in target lesion therapy | At the time of procedure
  Rate of change in treatment pattern from drug-eluting stents to drug-coated balloons in target lesion therapy
Cardiovascular death | 1 year
  Cardiovascular death
All-cause death | 1 year
  All-cause death
Non-fatal myocardial infarction (MI) | 1 year
  Non-fatal myocardial infarction (MI)
Target vessel MI excluding periprocedural MI | 1 year
  Target vessel MI excluding periprocedural MI
Target vessel MI including periprocedural MI | 1 year
  Target vessel MI including periprocedural MI
Clinically indicated target lesion revascularization | 1 year
  Clinically indicated target lesion revascularization
Clinically indicated target vessel revascularization | 1 year
  Clinically indicated target vessel revascularization
Any revascularization | 1 year
  Any revascularization
Vessel or stent thrombosis, definite or probable by Academic Research Consortium (ARC) definition | 1 year
  Vessel or stent thrombosis, definite or probable by Academic Research Consortium (ARC) definition
Cardiovascular death or target vessel MI | 1 year
  Cardiovascular death or target vessel MI
All-cause death or non-fatal MI | 1 year
  All-cause death or non-fatal MI
Target vessel failure (TVF), including cardiovascular death, target vessel MI, or clinically indicated target vessel revascularization | 1 year
  Target vessel failure (TVF), including cardiovascular death, target vessel MI, or clinically indicated target vessel revascularization
Target lesion failure (TLF), including cardiovascular death, target lesion MI, or clinically indicated target lesion revascularization | 1 year
  Target lesion failure (TLF), including cardiovascular death, target lesion MI, or clinically indicated target lesion revascularization
Cardiovascular death, target vessel MI, or vessel or stent thrombosis | 1 year
  Cardiovascular death, target vessel MI, or vessel or stent thrombosis
All-cause death, non-fatal MI, or clinically indicated target vessel revascularization | 1 year
  All-cause death, non-fatal MI, or clinically indicated target vessel revascularization
Major bleeding events (BARC type 2, 3, or 5) | 1 year
  Major bleeding events (BARC type 2, 3, or 5)

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Chair — +82-2-2072-2062
Locations (1):
- Bon-Kwon Koo, Seoul, South Korea